CLINICAL TRIAL: NCT06587815
Title: The Effect of a Musical Starry Sky Projector on Fatigue, Sleep, and Quality of Life in Pediatric Oncology Patients: A Randomized Controlled Trial Protocol
Brief Title: The Impact of a Musical Starry Sky Projector on Fatigue, Sleep, and Quality of Life in Pediatric Oncology Patients
Acronym: SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Associate Professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KOC UNI
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Oncology; Sleep Problems; Fatigue Intensity; Quality of Life
Keywords: fatigue, pediatric oncology, sleep, quality of life
MeSH Terms: conditions — Parasomnias; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Children in the control group were received standard care of the clinic
- Intervention Group (Experimental): Children in the intervention group received musical starry sky projector during the sleep time.
  Interventions: Other: musical starry sky projector

INTERVENTIONS:
Other: musical starry sky projector — Children in intervention group received musical starry sky projector during their sleep time
  Arms: Intervention Group

SUMMARY:
This study evaluated the effect of an Ocean Wave and LED Starry Sky Projector on fatigue, sleep, and quality of life in pediatric oncology patients.

DETAILED DESCRIPTION:
Sleep disturbances and fatigue were common issues among pediatric oncology patients, significantly impacting their overall quality of life. This study aimed to evaluate the effect of an Ocean Wave and LED Starry Sky Projector on fatigue, sleep patterns, and quality of life in this patient population. The research was structured as a parallel-group, randomized controlled trial. Pediatric oncology patients, aged 8-18 years, were recruited for participation.

The study intervention group used the Ocean Wave and LED Starry Sky Projector each night for one month, along with receiving the standard care typically provided in the oncology unit. The projector created a soothing visual and auditory environment designed to help induce relaxation, potentially improving sleep and reducing fatigue. Meanwhile, the control group received only the standard care offered to pediatric oncology patients, without the addition of the projector intervention. This study offered valuable insights into the use of non-pharmacological interventions for improving sleep quality and reducing fatigue among pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oncology patients aged 8-18 years.
* Recently diagnosed (< 1 month).
* Active receiving chemotherapy treatment
* Able to read and write in Turkish.
* Willing to participate voluntarily.

Exclusion Criteria:

* Being at the end of life
* Diagnosed with mental problems.
* Haemoglobin levels below 7 mg/dL).
* Having visual or hearing impairments.
* Unable to understand or communicate in Turkish.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Intensity Scale Score | It will be evaluated every day for one month.
  The FIS is an instrument developed to measure fatigue levels by Borneman et al., 2007. A single-item scale was created to measure fatigue intensity, rated on a scale from 0 to 10, where 0 represents no fatigue and 10 represents severe, overwhelming fatigue. The scale demonstrates face and content validity, with strong concurrent validity when compared to the Revised Piper Fatigue Scale and robust criterion validity. The scale relies on self-reporting by the patient, allowing for an accurate reflection of their fatigue levels. This tool will be administered daily throughout the intervention to monitor changes in fatigue levels (Borneman et al., 2007).
Visual Sleep Scale Score | It will be evaluated every day for one month.
  The primary outcome of this study will be to assess sleep quality and fatigue levels in pediatric oncology patients. The VSS is a visual tool designed to assess sleep quality in pediatric patients. The scale is scored from 1 to 10, with a higher score indicating poorer sleep quality. This scale offers a straightforward and intuitive method for evaluating the patient's perception of their sleep, making it suitable for use in a clinical setting.
Pediatric Quality of Life Inventory (PedsQL) Score | It will be evaluated every before the study and at the end of the first month.
  The PedsQL will be administered at two critical time points: at the baseline of the intervention and after one month. It is a validated tool for measuring health-related quality of life in children aged 2-18. It includes 23 items across four domains: physical health, emotional functioning, and social functioning, as defined by the World Health Organization. Additionally, it evaluates school functioning. The PedsQL provides three primary scores: Total Scale Score, Physical Health Summary Score, and Psychosocial Health Summary Score, derived from the emotional, social, and school functioning domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No